CLINICAL TRIAL: NCT05681780
Title: Clinical Trial of CD40L-augmented Tumor Infiltrating Lymphocytes (CD40L TIL) for Patients With Oncogene-Driven Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Clinical Trial of CD40L-Augmented TIL for Patients With EGFR, ALK, ROS1 or HER2-Driven NSCLC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21971
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Recurrent Non Small Cell Lung Cancer
Keywords: Lung Cancer; Tumor-Infiltrating Lymphocytes; EGFR Mutation; ALK Rearrangement; ROS1 Rearrangement; ERBB2 Mutation; HER2 Exon 20 Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Nivolumab; Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TIL+ Nivolumab (Experimental): Nivolumab infusion every 3 weeks prior to lymphodepletion chemotherapy with cyclophosphamide/fludarabine, TIL infusion and interleukin-2. Then nivolumab infusion every 4 weeks up to 12 months.
  Interventions: Biological: Tumor-infiltrating Lymphocytes (TIL); Drug: Nivolumab; Drug: Cyclophosphamide; Drug: Fludarabine; Other: Tumor-infiltrating Lymphocyte Therapy; Drug: Interleukin-2 (IL2)

INTERVENTIONS:
Biological: Tumor-infiltrating Lymphocytes (TIL) — Tumor harvest for TIL growth in the lab: A sample of the participant's tumor will be collected and sent to the lab for TIL growth. TIL will be prepared and cryopreserved.
  Other Names: TIL
Drug: Nivolumab — Nivolumab (Opdivo®), 360 mg, IV infusion every 3 weeks prior to TIL infusion, and then after TIL infusion 480 mg ever 4 weeks for up to 12 months.
  Other Names: Opdivo
Drug: Cyclophosphamide — Cyclophosphamide will be administered on days -7 and -6.
  Other Names: Cytoxan
Drug: Fludarabine — Fludarabine will then be infused per institutional standard on Days -7 to -3.
  Other Names: Fludara
Other: Tumor-infiltrating Lymphocyte Therapy — On day 0, all patients will receive a dose infusion TIL cells.
  Other Names: TIL
Drug: Interleukin-2 (IL2) — Participants will receive IL-2 for up to 6 doses, based on participants tolerance and investigator judgement. This will be given after the infusion of the T-cells.
  Other Names: IL2

SUMMARY:
To determine the effect of a special preparation of cells, called tumor-infiltrating lymphocytes (TIL) stimulated with CD40L, when given with the drug nivolumab, for patients with EGFR, ALK, ROS1, or HER2-genomically altered lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Diagnosis of stage IV or recurrent non-small cell lung cancer (NSCLC) with an activating genomic alteration within either: EGFR, ALK, ROS1, or ERBB2 receptor tyrosine kinase domains
* ECOG performance status of 0 or 1
* Expected survival ≥ 4 months
* Participants must have had disease progression after at least one prior line of systemic therapy for NSCLC, including appropriate prior targeted therapy for cases in which a targeted therapy is conventionally used for this genomic alteration, prior to initiating nivolumab trial therapy
* Measurable disease, not including any lesion that is used for TIL harvest, prior to initiation of nivolumab trial therapy
* In accordance with the criteria above, safely accessible tumor for TIL harvest by excisional biopsy expected to yield 1.5 cm3 of tissue, in aggregate
* Participants with known brain metastases are eligible for study enrollment if the brain metastases have received appropriate central nervous system-directed therapy or are found to be clinically stable ≤ 10 mm when comparing scans obtained during the screening period with a scan obtained ≥28 days prior, or if the treating physician determines that immediate CNS-specific treatment is not required prior to the first cycle of therapy. Please also refer to eligibility section on corticosteroids below.
* Adequate normal organ and marrow function as defined below:
* a. Hemoglobin ≥ 9.0 g/dL, with transfusions permissible;
* b. Absolute neutrophil count (ANC) ≥ 1000 per mm3);
* c. Platelet count ≥ 75,000 per mm3, without platelet transfusions for 7 days;
* d. Prothrombin Time ≤ 1.7x the institutional upper limit of normal (ULN), unless participant is receiving intended anticoagulant therapy.
* e. Serum bilirubin ≤ 2.0x the institutional ULN, or ≤ 4.0x ULN if confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology) with PI approval.
* f. AST/ALT ≤ 2.5x institutional ULN unless liver metastases are present, in which case it must be ≤ 5x ULN
* g. Serum creatinine of ≤ 1.5x institutional ULN, or ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* h. Albumin ≥ 2.0 g/dl
* Pulmonary function tests within past 4 months showing DLCO ≥45% of predicted. Adjusted DLCO based on hemoglobin concentration should be used, if available.
* Human immunodeficiency virus (HIV)-infected participants must be receiving on effective antiretroviral therapy for past 6 months with undetectable viral load and normal CD4 count
* Participants with history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy, if indicated, and no overt cirrhosis
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they must have an undetectable HCV viral load and no overt cirrhosis
* Participants with a prior or concurrent malignancy must have a natural history which does not have the potential to interfere with safety or efficacy assessment of the investigational regimen

Exclusion Criteria:

* No more than six prior lines of systemic therapy for NSCLC
* No prior PD-1 or PD-L1 inhibitor treatment for metastatic NSCLC. Examples of inhibitors include: nivolumab, atezolizumab, pembrolizumab, avelumab, cemplimumab, spartalizumab, or durvalumab.
* Participants with rapidly progressing tumors, as judged by the investigator
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, limited site eczema, or limited site plaque psoriasis not requiring systemic treatment (within the past 2 years), or other autoimmune conditions which are not expected to recur, are allowed after approval from the medical monitor or PI
* Active leptomeningeal or pachymeningeal metastases, or carcinomatous meningitis. This is due to prognostic implications and timeline for cell therapy
* Has a diagnosis of primary immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* a. Oral hydrocortisone, only for the purposes of a documented adrenal insufficiency diagnosis, is permitted if ≤ 25 mg daily total dose
* b. Inhaled, intranasal, or topical corticosteroids are permitted
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than atrial fibrillation or supraventricular tachycardia), and significant ≥85% carotid artery stenosis
* Unresolved toxicity (grade 2) from previous anti-cancer therapy. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripheral neuropathy)
* Mean QT interval corrected for heart rate (QTc) ≥480 ms calculated from electrocardiograms (EKGs) using Bazett's Correction
* Participants with active systemic infections requiring intravenous antibiotics within 1 week prior to nivolumab. Prophylactic, empiric, or suppressive antibiotics are permitted with sponsor approval
* History of allogeneic organ transplant
* Participants with psychiatric illness/social situations that would limit compliance with study requirements
* Participants with a history of anaphylaxis to beta-lactam antibiotics. Patients may be evaluated for reported history by conducting a history and physical, and a skin test/challenge where appropriate under medical guidance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to 18 Months
  To characterize the safety profile of CD40L-augmented TIL administered with nivolumab.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 5 Years
  Proportion of patients with complete response + partial response (CR+PR) per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Duration of Response (DOR) | Up to 5 years
  The time from the date of the first documentation of initial response (CR or PR) to the date of the first documentation of progressive disease (PD) or death due to any cause.
Overall Survival (OS) | Up to 5 Years
  The time length of patients living from the date of TIL infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ben Creelan, MD, MS, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Creelan BC, Wang C, Teer JK, Toloza EM, Yao J, Kim S, Landin AM, Mullinax JE, Saller JJ, Saltos AN, Noyes DR, Montoya LB, Curry W, Pilon-Thomas SA, Chiappori AA, Tanvetyanon T, Kaye FJ, Thompson ZJ, Yoder SJ, Fang B, Koomen JM, Sarnaik AA, Chen DT, Conejo-Garcia JR, Haura EB, Antonia SJ. Tumor-infiltrating lymphocyte treatment for anti-PD-1-resistant metastatic lung cancer: a phase 1 trial. Nat Med. 2021 Aug;27(8):1410-1418. doi: 10.1038/s41591-021-01462-y. Epub 2021 Aug 12. PMID 34385708
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=21971